CLINICAL TRIAL: NCT07023185
Title: Cold and Compression After Total Knee Arthroplasty for Pain Attenuation: A Randomized, Controlled Trial
Brief Title: Cold and Compression Post TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: BREG, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025.069
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Primary Osteoarthritis Patients Scheduled for Total Knee Replacement Surgery
Keywords: total knee replacement; primary osteoarthritis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care Arm (Active Comparator): Patients in this arm will receive standard therapy post-surgery and discharged with 28 hydrocodone/APAP 7.5 mg pills taken every 6 hours as needed (or its MME equivalent), 1 identical refill if patient calls, and cold therapy (bag of ice or gel pack)
  Interventions: Other: SOC (Standard of care)
- Cold and Compression (Experimental): Patients in this arm will be discharged with 28 hydrocodone/APAP 7.5 mg pills taken every 6 hours as needed (or its MME equivalent), 1 identical refill if patient calls, and cold & compression therapy device provided by Sponsor)
  Interventions: Device: Cold and Compression

INTERVENTIONS:
Device: Cold and Compression — External mechanical compression therapy (e.g., compression stockings) has been shown to reduce swelling and risk of deep vein thrombosis in the lower limbs following TKA.12,13 Combining advanced cryotherapy (continuous circulating cold flow) and dynamic compression may offer added benefits than either traditional cryotherapy (e.g., cold packs) or compression (e.g., stockings) alone.
  Arms: Cold and Compression
Other: SOC (Standard of care) — Patients enrolled in this arm will be discharged with 28 hydrocodone/APAP 7.5 mg pills taken every 6 hours as needed (or its MME equivalent), 1 identical refill if patient calls, and cold therapy (bag of ice or gel pack)
  Arms: Standard of Care Arm

SUMMARY:
The purpose of this study is to compare pain score (Patient-Reported Outcomes Measurement Information System: PROMIS NRS Pain Subscale) between the control and cold/compression groups pre-surgically, daily after surgery for 14 days, then weekly after surgery for 3 months, and at 6 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 yr or older
2. Patient of Dr. Howard Hirsch or Dr. Vinod Dasa scheduled for total knee arthroplasty (knee replacement) at Ochsner Kenner
3. Will receive outpatient physical therapy at OTW Driftwood for the entire post-op rehabilitation period
4. English speaking
5. Diagnosis of primary osteoarthritis

Exclusion Criteria:

1. Chronic opioid use
2. Opioid use within the last 3 months
3. PCS score ≥ 30
4. Diagnosis of inflammatory disease process (i.e., gout, rheumatoid arthritis, systematic lupus erythematosus...)
5. Discharge to skilled nursing
6. Cold intolerance related to diseases, like Raynaud's
7. Significant vascular impairment in the affected region
8. Current clinical signs of inflammatory phlebitis, venous ulcers, or cellulitis
9. Significant risk factors or current clinical signs of embolism (e.g., pulmonary embolus, pulmonary edema, cerebral infarction, atrial fibrillation, endocarditis, myocardial infarction, or atheromatous embolic plaque)
10. A condition in which increased venous or lymphatic return is not desired in the affected extremity (e.g., lymphedema after breast cancer or other local carcinoma and/or carcinoma metastasis in the affected extremity).
11. Uncontrolled hypertension (physician discretion), cardiac failure, extreme low blood pressure, or decompensated cardiac insufficiency.
12. Localized unstable skin condition (e.g., dermatitis, vein ligation, gangrene, or recent skin graft) in the affected region.
13. Had recent toe surgery in the affected region
14. Current clinical signs in the affected region of significant peripheral edema (e.g., deep vein thrombosis, chronic venous insufficiency, acute compartment syndrome, systemic venous hypertension, congestive heart failure, cirrhosis/liver failure, renal failure).
15. An acute, unstable (untreated) fracture in the affected region.
16. Any active local or systemic infection.
17. Obtunded or with diabetes mellitus, multiple sclerosis, poor circulation, spinal cord injuries, and rheumatoid arthritis
18. Areas of skin breakdown or damage (damaged or at-risk skin) producing uneven heat conduction across the skin (e.g., open wound, scar tissue, burn or skin graft). Any open wound must be dressed prior to use of the Polar Care Wave System.
19. Presumptive evidence of congestive heart failure
20. Pre-existing DVT condition
21. Deep acute venal thrombosis (Phlebothrombosis)
22. Episodes of pulmonary embolism
23. Pulmonary edema
24. Acute inflammation of the veins (Thrombophlebitis)
25. Decompensated cardiac insufficiency
26. Arterial dysregulation
27. Erysipelas
28. Carcinoma and carcinoma metastasis in the affected extremity
29. Decompensated hypertonia
30. Acute inflammatory skin diseases or infection
31. Venous or arterial occlusive disease
32. Medical situations where increased venous or lymphatic return is undesirable
33. Poor peripheral circulation
34. Severe arteriosclerosis, or active infection
35. Known hematological dyscrasias that predispose to thrombosis (e.g., paroxysmal cold hemoglobinuria, cryoglobulinemia, sicklecell disease, serum cold agglutinins).
36. Tissues inflamed as a result of recent injury or exacerbation of chronic inflammatory condition.
37. Compromised local circulation or neurologic impairment (including paralysis or localized compromise due to multiple surgical procedures or diabetes) in the affected region.
38. Cognition or communication impairments that prevent them from giving accurate and timely feedback.
39. Cold allergy
40. Cold agglutinin disorders like paroxysmal cold hemoglobinuria
41. Buerger's disease
42. Chilblains
43. Cryoglobulinemia
44. Sickle cell anemia
45. Uncontrolled diabetes (physician discretion)
46. Hypersensitivity to cold
47. History of cold injury
48. Severe cardiovascular disease, anesthetic skin, hypercoagulation disorders, poor circulation, extremities sensitive to pain, extremely low blood pressure that are incapacitated, decreased skin sensitivity, vein ligation or recent skin grafts, or pheochromocytoma.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
PROMIS Pain NRS subscale | Enrollment to 6 months post-surgery
  Compare pain score (Patient-Reported Outcomes Measurement Information System: PROMIS NRS Pain Subscale) between the control and cold/compression groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Medical Center - Kenner, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Currently there are no plans to share the data as there are no data sharing agreements in place with other institutions.